CLINICAL TRIAL: NCT01003470
Title: Treating Apoplectic Sequela With Acupuncture: a Randomized Controlled Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Ministry of Science and Technology of the People's Republic of China, State Administration of Traditional Chinese Medicine of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTRDP- 2006BAI12B02-2
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Cerebral Infarction
Keywords: cerebral infarction; Paralysis; acupuncture; rehabilitation; trial
MeSH Terms: conditions — Cerebral Infarction; Paralysis | interventions — Acupuncture Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- acupuncture (Experimental)
  Interventions: Other: acupuncture
- rehabilitation (Active Comparator)
  Interventions: Behavioral: rehabilitation
- acupuncture and rehabilitation (Active Comparator)
  Interventions: Other: acupuncture and rehabilitation

INTERVENTIONS:
Other: acupuncture — Xing Nao Kai Qiao Acupuncture
  Arms: acupuncture
Behavioral: rehabilitation — Kinesitherapy
  Arms: rehabilitation
Other: acupuncture and rehabilitation — Xing Nao Kai Qiao Acupuncture plus Kinesitherapy
  Arms: acupuncture and rehabilitation

SUMMARY:
The purpose of this study is to evaluate the therapeutic effect of acupuncture method of "Xing Nao Kai Qiao" for paralysis as an apoplectic sequela in a multicenter randomized and controlled clinical trial and to compare the efficacy between acupuncture and rehabilitation therapy. In addition, evaluating the trial in the view of medical economics.

DETAILED DESCRIPTION:
This study is a multi-center randomized controlled trial comparing three treatment groups.The trial is completed in the following three hospitals: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (TCM) of China, Tianjin Hospital of TCM of China, and Qingdao Haici Medical group of Shangdong province of China.

The total observation period within this study is 24 weeks for each patient. All patients should remain hemiplegia within 15～90 days after stroke. After randomization the patients will receive 4 sessions of 30 minutes' duration during a period of 4 weeks. The outcome measurement is completed both in the different times as follows: before treatment, after the first treatment, 7, 14, 28days after treatment and follow up at 6 months after treatment.

288 patients were randomised into three groups: acupuncture group, rehabilitation group,and acupuncture plus rehabilitation group.The patients in the three groups are blinded as to which treatment method they received. The central randomization is used in this trial, which is performed by the Drug Clinical Research Center of Shanghai University of TCM of China. This trial is performed according to the principles of the Declaration of Helsinki (Version Edinburgh 2000). And the trial protocol has been approved by local institutional review board and ethics committee.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral infarction diagnosed according to the diagnostic standard of western medicine
2. Apoplexy diagnosed according to the diagnostic standard of traditional Chinese medicine for apoplexy
3. Cerebral vascular accident occured in the internal carotid artery system which was verified by cerebral CT or MRI
4. The incidence of apoplexy less than twice and the time of onset 15~3 months
5. Age: 40-75 years, non-limited gender
6. NDS score of limb functional defect ≥10
7. The patient was alert and the vital signs are stable
8. Participant signed the informed consent form

Exclusion Criteria:

1. TIA or RIND
2. The nerve function defect induced by the cerebral tumor, trauma, parasitic diseases, heart disease and metabolic disorder or hemorrhagic cerebrovascular disease
3. Pregnant or breast-feeding women
4. Complicated with severe primary disease in heart, liver, kidney and hematology system or psychopath

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Score of neurological defect | before treatment, after the first treatment, 7, 14, 28days after treatment and follow up at 6 months after treatment.

SECONDARY OUTCOMES:
Visualized anologue score | before treatment, after the first treatment, 7, 14, 28days after treatment and follow up at 6 months after treatment.
Spasm evaluation | before treatment, after the first treatment, 7, 14, 28days after treatment and follow up at 6 months after treatment.
Safety evaluation | before treatment, after the first treatment, 7, 14, 28days after treatment and follow up at 6 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sicheng Wang, Master, Study Director — State Administration of Traditional Chinese Medicine of China
Locations (1):
- First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (TCM), Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Shiflett SC. Does acupuncture work for stroke rehabilitation: what do recent clinical trials really show? Top Stroke Rehabil. 2007 Jul-Aug;14(4):40-58. doi: 10.1310/tsr1404-40. PMID 17698457
- See also: Related Info — http://www.most.gov.cn/